CLINICAL TRIAL: NCT07038603
Title: Assessing the Feasibility of Behavioural Activation (BA) to Support People With Parkinson's Disease Enhanced by a Virtual Reality Exercise Programme
Brief Title: Feasibility of a Behavioural Activation Protocol to Support People With Parkinson's Enhanced by VR
Acronym: BAPP-VR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University, Belfast (Other)
Collaborators: Marie Curie Hospice, Belfast (Other); Parkinson's UK (Other)
Responsible Party: Principal Investigator, Dr Paul Best, Principal Investigator, Queen's University, Belfast
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: B22/27
Record Dates: First submitted 2024-02-19; First posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Parkinson Disease
Keywords: anxiety; depression
MeSH Terms: conditions — Parkinson Disease; Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: The single group study is a small-scale feasibility study using a pre-test and post-test design. All participants will receive the same/ adapted Behavioural Activation (BA) protocol and Virtual Reality exercise programme.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Behavioural Activation enhanced by Virtual Reality exercises (Experimental): Participants will attend a 6 week BA group talking therapy (50mins-1hour) followed by a (30 min) exercise session enhanced with the use of Virtual Reality. Participants will be immersed in a virtual reality forest where they will complete a variety of physio chosen exercises. This intervention will be run in three phases.
  Interventions: Other: BAPP-VR

INTERVENTIONS:
Other: BAPP-VR — A carefully considered adaptation of a BA protocol enhanced with the use of VR

SUMMARY:
The proposed research project will involve developing and testing the feasibility of a 6 week Behavioural Activation (BA) programme for people with Parkinson's Disease, which will be enhanced by Virtual Reality exercise programme. The aim of the programme will be to support the mental well-being and physical rehabilitation of people with Parkinson's Disease who are known to Marie Curie Outpatient Department (Belfast).

The main question[s] it aims to answer are:

Is a Behavioural Activation (BA) enhanced by a Virtual Reality exercise programme feasible and can it support the mental well-being and physical rehabilitation of People with Parkinson's Disease ?

Can the potential impacts of the intervention help to reduce anxiety and depression, as well as improve balance, social interaction and adherence to the programme?

Participants will:

* Attend a group for 6 weeks with the addition of an introductory session, for 1.5 hours per session.
* During sessions they will be asked to take part in a Behavioural Activation talking therapy. The aim of the intervention is to engage patients through activation strategies and help support adherence to exercise programmes. Participants will complete 'homework' tasks between sessions.
* In addition to this, the BA intervention will be enhanced by Virtual Reality exercises and participants will complete exercises within the immersive space using a VR headset.
* Data collection will capture any changes in depression, anxiety, balance,social interaction and adherence to the programme.
* The intervention will be carried out in three phases.

DETAILED DESCRIPTION:
The research design will be a small-scale feasibility study. The study will use a pre-test and post-test design to assess the feasibility of Behavioural Activation (BA) to support people with Parkinson's Disease enhanced by a Virtual Reality exercise programme.

Aims and objectives:

This research aims to address this gap in the evidence base by developing and testing the feasibility of a Behavioural Activation (BA) enhanced by a Virtual Reality exercise programme for supporting the mental well-being and physical rehabilitation of People with Parkinson's Disease.

1. Developing and creating a Behavioural Activation intervention
2. Determine recruitment and retention rates
3. Test the feasibility of Behavioural Activation (BA) enhanced by Virtual Reality exercise for people with Parkinson' s Disease.
4. Pilot technology and methodological procedures
5. Explore the potential impacts of the intervention in reducing anxiety and depression, as well as improving balance, social interaction and adherence to the programme.

The study will be conducted under the supervision of the senior Physiotherapist, another physiotherapist and research nurse at the recruiting hospice site, alongside the researcher and other designated members of the clinical team. The intervention will take place in both the clinical setting at the hospice, as well as in the domiciliary setting. Quantitative data will be collected via pre and post-test outcome measures. Qualitative data will supplement findings to assess the acceptability of the intervention, frequency of use, as well as motivation, ease of use within the home setting, adaptation and adherence.

Primary Outcomes:

To test the feasibility of Behavioural Activation (BA) to support people with Parkinson's Disease enhanced by a Virtual Reality exercise programme.

Secondary Outcomes:

The potential benefits of BA enhanced by a Virtual Reality exercise-based programme in reducing depression, anxiety and improving balance, social interaction and adherence to the programme.

Intervention :

Introductory Sessions, training and baseline outcomes The intervention will replace a 6-week rehabilitative exercise intervention programme at the clinic with the addition of BA. Baselines measures will be taken at the introductory session by the senior physiotherapist and/or physio team.

BA intervention led initially by psychotherapist enhanced by VR Participants will complete the 6-week Behaviour Activation BA programme led by the Doctorate of Philosopy (PhD) researcher who is a qualified psychotherapist (British Association of Behavioural & Cognitive psychotherapies BABCP). Previous VR exercise studies have used a variety of durations and frequencies for similar interventions. The researcher has followed the clinical advice of the head physiotherapist to determine the duration of the intervention in this study. The intervention is a concise and carefully adapted Behavioural Activation for depression treatment protocol by Elkers and Dawson The group sessions will last for 1.5 hours, examples see listed below. Each session will have a psycho-educational element, such as behaviour/mood link (session 2) This session will support participants to create a problems list and consider setting personal goals. As an introduction to VR, participants will have the opportunity to trial out the Cognitive Behavioural Therapy (CBT) relaxation immersive scene during the class. Any issues with technology or practicalities can be discussed plus patients can share initial experiences of use. Participants will be asked to complete 'homework' between sessions and build in the VR exercise element into the structure of their week, this will become progressively more intense as sessions develop. Patients will also receive a pack of resource worksheets for the BA programme sent via email or participants can request a paper copy. The structure is informed by a current online and in-clinic conventional programme delivery run by Marie Curie.

The researcher will carry out the research in three - phases:

Phase 1: Literature Review and intervention development Phase 2: First group intervention (6 participants) Phase 3: Second, third and fourth group intervention ( larger cohort 14 -18 participants - this may be run as 3 separate groups. More refined based on reflection of Phase 2 )

Steps to participant journey:

Step 1: Participants will have the opportunity to receive guidance on the use of the VR equipment (Oculus Quest), as well as being provided with a written and video resource to take home at an introductory session at the Marie Curie Clinic. Pre-test baseline measures will also be taken during this session by qualified psychotherapist. Consent will also be taken. Cares and Healthcare Professionals will also be invited to this session.

Step 2: Patients will meet in a weekly group in person at the Marie Curie Clinic. The Agenda will allow for group discussion/support, Psycho-education BA strategies, training and implementation of VR to enhance the programme and homework setting and reflection. Patients will be encouraged to set goals between sessions and to complete homework using a combination of resources and exercises as well as CBT relaxation techniques.

There are 4 main exercises which encourage patients to use upper and lower limb mobility. To give an example, one of the exercises requires the patient to use upper limb movements to reach and select changing coloured dots. Patients are encouraged to improve their scores as they progress. The setting of the exercise is in an immersive forest scene. VR interventions will be set up and carefully considered, goal orientated and reflected upon weekly.

Step 3: Participants will be invited to take part in semi-structured interviews via Microsoft Teams or phone-call, as well as complete questionnaire and complete post-test outcome measures. Healthcare professionals and carers will be asked to take part in semi-structured interviews to gain their perspective on the intervention.

Study Setting:

Participants will be recruited from the Parkinson's clinic based at Marie Curie, Belfast and through advertising at Parkinson's UK. The clinic offers outpatient physiotherapy support to people with Parkinson's in Northern Ireland. The study will take place at the Marie Curie Clinic.

Participants:

Participants will have a diagnosis of Idiopathic Parkinson's Disease and carers and healthcare staff will also be recruited to gain their perspective on the project.

Recruitment:

Parkinson's UK are advertising for the study in order to meet the recruitment numbers required and acting as the gatekeeper.

After ethical approval a member of the research team will offer a Participant Information Sheet (PIS) to patient, carers and healthcare staff. Patients will be allowed at least 48 hours to consider participation, prior to being asked if they verbally consent to participate.

The physio team will arrange a screening for the inclusion criteria re. physical outcomes.

A member of the research team will call the participant to kindly answer some pre-intervention questions. Once included they will be invited to an introductory session. The research team will also ask the participant to discuss if their carer may be open to attending the introductory session and they will be provided with a PIS and they too will be given 48 hours to verbal consent before being contacted by a member of the research team. Written consent will be given at the introductory session.

Analytical methods and Evaluation

Primary outcomes:

The feasibility of Behavioural Activation (BA) to support people with Parkinson's Disease enhanced by a Virtual Reality exercise programme.

Quantitative data will be analysed to evaluate recruitment and retention capacity. Qualitative data will further inform reasons for drop out rates, acceptability of outcomes measures determined by patient feedback on the level of burden to complete questionnaires, at pre-post data collection, along with monitoring of how many questionnaires are completed and reasons for non-completion. Qualitative data will be managed using the Nvivo V.11 software.

Questionnaires will be distributed to evaluate the acceptability and suitability of the BA intervention enhanced by the Virtual Reality exercise programme, as well use of the VR element and delivery of BA via telecommunication. Semi-structured interviews will also be carried out with patients, carers and physiotherapists involved in the project to evaluate participant response to the intervention. Follow up questions will be evaluated to consider barriers and success of the research and revision made for Phase 3 and 4. Interviews will be digitally recorded. Recordings will be deleted following transcription, and all identifying information will be removed from the transcripts to ensure participant anonymity.

Written informed consent will be secured prior to commencing semi-structured interviews. An experienced qualitative researcher will interview participants to ensure rigour. Interviews will take place via Microsoft Teams for a duration of 45 minutes. Data will be analysed by the researcher using a thematic content analysis. Nvivo V.11 software will be used to manage qualitative data.

Secondary Outcomes:

Baseline measures will be provided to participants during the introductory session. Physical outcomes measures (Berg Balance Scale) will be completed as well as, anxiety (GAD-7) and depression measures Patient Health Questionnaire (PHQ-9). Secondary outcomes will be analysed and evaluated using the Statistical Package for Social Sciences, v20. As this is a feasibility study there is no formal power calculation. Confidence intervals will be provided along with any estimates, and any change in outcome scores between baseline (prior to the intervention), and post intervention outcomes. Adherence rates will also be analysed and evaluated post intervention.

Quantitative data using outcome measures; Berg Balance Scale, PHQ-9 and GAD-7 will be collected pre and post-test, as well as recruitment (number of participants at the beginning of the study) and retention (numbers that complete the study).

Descriptive statistics including means and standard deviations will be gathered at each time point for each outcome.

Feasibility will be assessed using anxiety and depression as well as balance outcomes; ability to recruit and retain; and fidelity (i.e. consistency of implementation across groups). Acceptability will be assessed by comparing attendance across groups, dropout rates and using through the qualitative methods (interviews and observations) specified to explore (1) reasons for taking part; and (2) user satisfaction.

The quantitative data will be analysed using the Statistical Package for Social Sciences (SPSS), version 25.0 software.

Semi-structured interviews and focus groups will be carried out and evaluated to determine the acceptability and suitability of the BA intervention on secondary outcomes; physical, anxiety and depression, social interaction and adherence. Semi-structured interviews will also be carried out with patients, carers and physiotherapists involved in the project to evaluate participant response to secondary outcomes. Interviews will be digitally recorded. Recordings will be deleted following transcription, and all identifying information will be removed from the transcripts to ensure participant anonymity.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of Idiopathic Parkinson's Disease which has been diagnosed by a neurologist.
* Patients with an early to moderate disease stage Hoehn and Yahr scale 1-3
* Patients with a BERG Balance Scale > 45
* Currently not attending any other rehab programme/participation in another clinical trial
* Able to exercise independently & mobilise
* No hospitalisation or medication change within the past month
* No other serious medical or surgical condition

Carers:

• Have direct contact with a participant on the BAPP-VR programme in the role of a carer.

Healthcare staff:

• Have helped in some capacity to facilitate the intervention or referred patients to BAPP-VR

Exclusion Criteria:

* Those who are unwilling/unable to provide written consent to participate
* Not receiving another form of psychotherapy
* Actively suicidal
* No other Neurological Condition
* Vision/ auditory impairment.

Carers and healthcare staff:

• Those who are unwilling/unable to provide written consent to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2023-04-05 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
GAD-7 | From enrolment to the end of treatment - week 6
  Anxiety Measure - lower score better outcome - out of possible score of 21
Berg Balance Scale | From enrolment to the end of treatment - week 6
  Balance test - higher score better outcome - out of possible score of 56
PHQ-9 | From enrolment to the end of treatment - week 6
  Derpession measure - lower score better outcome -out of possible score of 27

CONTACTS AND LOCATIONS:
Overall Officials: Paul Best, Reader, Principal Investigator — Queen's University, Belfast
Locations (1):
- Marie Curie, Belfast, United Kingdom

IPD SHARING:
Plan to Share IPD: No